CLINICAL TRIAL: NCT07260942
Title: Ferroptosis Role in the Pathophysiology of Systemic Lupus Erythematosus
Acronym: FERROLUP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2025/003
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; ferroptosis; autoimmunity
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic lupus erythematosus (SLE) (Experimental)
  Interventions: Biological: blood sample
- Rheumatoid arthritis or an inflammatory bowel (Active Comparator)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — 30 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation

SUMMARY:
The study aims at defining the role of ferroptosis s in the physiopathology of systemic lupus erythematosus (SLE). Ferroptosis (phenomenon of cellular death regulated by iron) is a metabolic pathway potentially implicated in SLE with potential for the discovery of new therapeutic strategies.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a complex autoimmune disease affecting various organs. Regulatory T cells (Treg) and platelets play a crucial role in the pathogenesis of SLE by regulating immunity and promoting inflammation. Ferroptosis, an iron-regulated cell death process, is emerging as a key player in many diseases, including SLE.

The project, FERROLUP, aims to understand the role of ferroptosis in SLE and to explore the therapeutic potential of selenium compounds to modulate this process. Recent work has identified down-regulation of glutathione peroxidase 4 (GPx4) by immune complexes and interferon-alpha in neutrophils, leading to ferroptosis and worsening of SLE. In addition, data suggest the involvement of ferroptosis in lupus nephritis.

The Bordeaux team has developed selenium compounds, GPx4 mimics, capable of inhibiting ferroptosis in lupus neutrophils. These compounds have shown promising efficacy in mouse models and preliminary human studies in another inflammatory disease. The FERROLUP project aims to characterize the level of lipid peroxidation and GPx4 expression in SLE patients, and to test the impact of selenium compounds on the inhibition of ferroptosis induced by P-selectin, a molecule involved in Treg dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* diagnosis of systemic lupus erythematosus;
* being affiliated to health insurance, willing to participate and to sign informed consent;
* control group : patients with a diagnosis of rheumatoid arthritis or an inflammatory bowel disease.

Exclusion Criteria:

* pregnant or breastfeeding women;
* patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of lipid peroxidation in regulatory T lymphocytes population in lupus subjects. | At baseline (Day 0)

SECONDARY OUTCOMES:
Measurement of lipid peroxidation in regulatory T lymphocytes population in lupus subjects and controls. | At baseline (Day 0)
Measurement of lipid peroxidation in other immune cells (T and B lymphocyte populations) in lupus subjects and controls | At baseline (Day 0)
GPX4 expression in lupus subjects and controls. | At baseline (Day 0)
Correlation between ferroptosis markers and the level of activity in B lymphocyte populations | At baseline (Day 0)
In-vitro effect of BXT on different T lymphocytes population in the presence of P-selectin in sera of lupus subjects and controls | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe RICHEZ, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de rhumatologie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No